CLINICAL TRIAL: NCT02573688
Title: Interdisciplinary Intervention Project - Promotion and Rehabilitation in Patients With Obesity and Other Metabolic Diseases
Brief Title: Interdisciplinary Intervention in Patients With Obesity and Other Metabolic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Danielle Arisa Caranti, PhD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIDM-2014-GEO
Record Dates: First submitted 2015-10-02; First posted 2015-10-12 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Obesity
Keywords: Obesity; Metabolic Syndrome X; Interdisciplinary Studies
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interdisciplinary Therapy (Experimental): The Therapy includes: Physical Exercise (three times week - 180 minutes); Nutrition, Psychology, Physiotherapy (once a week - 60 minutes each one)
  Interventions: Behavioral: Interdisciplinary Therapy

INTERVENTIONS:
Behavioral: Interdisciplinary Therapy — The nutrition intervention will consist of group meetings and prescription of individual diets. Participants will have dietary lessons, with information related to the improvement of food consumption and nutritional quality. Exercise program will be focused on improving activity habits, leading to increased energy expenditure. They will undergo training sessions containing aerobic and resistance training. In Psychological program, participants will be monitored in the support group and, if necessary, individual psychological therapy is recommended. The sessions will discuss common psychological aspects commonly associated with obesity (depression, anxiety, stress, family problems, body image, eating disorders and others). The physiotherapy interventions aim to increase functional capacity.
  Other Names: Obesity Treatment; Lifestyle Improvement

SUMMARY:
The aim of the research study will be assess the effectiveness of a long-term interdisciplinary lifestyle in many aspects including food intake, psychological symptoms, physical activity habits, energy expenditure, body composition and anthropometric measurements in adults obese.

DETAILED DESCRIPTION:
Participants will be recruited after dissemination of the program in the local media and internet.

They will go through a short interview to evaluate inclusion and exclusion criteria. Thus, all obese adults will be submitted to an interdisciplinary lifestyle modification therapy according the inclusion criteria.

The interdisciplinary therapy will consist of nutritional, physical exercise, psychological and physiotherapy support during the course of one year, according the literature the investigators promote a long term therapy to control obesity and metabolic diseases.

The participants will be evaluated at baseline and after the therapy in accordance with Ethical guidelines.

The main purpose of this therapy is to enhance the quality of life of the participants promoting an active lifestyle and quality of life, adherence a healthy nutritional habits and a healthy weight loss.

Our focus will be on teaching strategies to maintain a healthy life style behaviors after therapy, our protocol is in agreement with public health field in this way.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 50 years and body mass index (BMI) between 30 and 39.9 Kg/m2

Exclusion Criteria:

* Musculoskeletal limitations preventing the practice of physical exercise, other metabolic or endocrine diseases, identified genetic diseases, pregnancy, previous drug utilization and excessive chronic alcohol consumption

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Body Mass | one year
  Body Mass (kg)
Physical Activity | one year
  Quadrimensional accelerometer

SECONDARY OUTCOMES:
Total Cholesterol. | one year
  Blood lipid fraction (mg/dL) after 12h overnight fasting.
High Density Lipoprotein - Cholesterol | one year
  HDL-c; Blood lipid fraction (mg/dL) after 12h overnight fasting.
Triglycerides | one year
  Blood lipid fraction (mg/dL) after 12h overnight fasting.
Glucose levels. | one year
  Glucose levels (mg/dL) after 12h overnight fasting.
Waist circumference | one year
  Anthropometric measure (cm)
Blood Pressure | one year
  Systolic and Diastolic Blood pressure (mmHg)
Improvement in Quality of Life | One year
  WHO - Quality of life Brief Questionnaire
Cardiorespiratory parameters | One year
  Maximal ergometer test. Maximal oxygen uptake.
Resting Metabolic Rate | One year
  Indirect calorimetry test (kcal/day)
Psychological Parameters - Anxiety | one year
  Anxiety, Beck´s Anxiety Inventory Questionnaire (Score)
Psychological Parameters - Depression | one year
  Depression; Beck´s Depression Inventory Questionnaire (Score)
Physiotherapy parameters | one year
  Functional capacity - Health Assessment Questionnaire (Score)
Nutritional parameters | one year
  Macronutrient, micronutrient and calorie intakes
Inflammatory markers | one year
  adipokines status

CONTACTS AND LOCATIONS:
Overall Officials: Danielle A Caranti, PhD, Study Director — Federal University of São Paulo
Locations (1):
- GEO - Obesity Study Group, Santos, São Paulo, Brazil

REFERENCES:
- [Background] Jamar G, Pisani LP, Medeiros A, Oyama LM, Masquio DC, Colantonio E, Garcia S, Sanches RB, dos Santos Moraes A, Belote C, Caranti DA. Effect of Fat Intake on the Inflammatory Process and Cardiometabolic Risk in Obesity After Interdisciplinary Therapy. Horm Metab Res. 2016 Feb;48(2):106-11. doi: 10.1055/s-0035-1548871. Epub 2015 Sep 15. PMID 26372897
- [Background] Moraes Ados S, Pisani LP, Corgosinho FC, Carvalho LO, Masquio DC, Jamar G, Sanches RB, Oyama LM, Damaso AR, Belote C, Caranti DA. The role of leptinemia state as a mediator of inflammation in obese adults. Horm Metab Res. 2013 Aug;45(8):605-10. doi: 10.1055/s-0033-1343450. Epub 2013 May 13. PMID 23670346
- [Background] Jamar G, Pisani LP, Oyama LM, Belote C, Masquio DC, Furuya VA, Carvalho-Ferreira JP, Andrade-Silva SG, Damaso AR, Caranti DA. Is the neck circumference an emergent predictor for inflammatory status in obese adults? Int J Clin Pract. 2013 Mar;67(3):217-24. doi: 10.1111/ijcp.12041. PMID 23409690
- [Background] Carvalho-Ferreira JP, Cipullo MA, Caranti DA, Masquio DC, Andrade-Silva SG, Pisani LP, Damaso AR. Interdisciplinary lifestyle therapy improves binge eating symptoms and body image dissatisfaction in Brazilian obese adults. Trends Psychiatry Psychother. 2012;34(4):223-33. doi: 10.1590/s2237-60892012000400008. PMID 25923071
- [Background] Sanches RB, Andrade-Silva SG, Rossi S, Fidalgo JPN, Moraes AS, Jamar GGQ, Colantonio E, Botero JP, dos Santos RVT, Caranti DA. Body composition and aerobic fitness in obese women: beneficial effects of interdisciplinary therapy. Brazilian Journal of Physical Activity and Health 18(3):354-362, 2013
- [Derived] Moraes ADS, Padovani RDC, La Scala Teixeira CV, Cuesta MGS, Gil SDS, de Paula B, Dos Santos GM, Goncalves RT, Damaso AR, Oyama LM, Gomes RJ, Caranti DA. Cognitive Behavioral Approach to Treat Obesity: A Randomized Clinical Trial. Front Nutr. 2021 Feb 18;8:611217. doi: 10.3389/fnut.2021.611217. eCollection 2021. PMID 33681273